CLINICAL TRIAL: NCT00457249
Title: Safety and Immunogenicity of Tetanus Toxoid, Reduced Diphtheria Toxoid and Acellular Pertussis Vaccine Adsorbed (ADACEL®) in Persons ≥65 Years of Age
Brief Title: A Trial to Evaluate the Safety and Immunogenicity of ADACEL® Vaccine in Persons 65 Years of Age and Older
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: TD515
Record Dates: First submitted 2007-04-05; First posted 2007-04-06 (Estimated); Results first posted 2012-10-19 (Estimated); Last update posted 2012-10-19 (Estimated); Status verified 2012-09

CONDITIONS: Pertussis; Tetanus; Diphtheria
Keywords: Pertussis; Tetanus; Diphtheria; Tdap
MeSH Terms: conditions — Whooping Cough; Tetanus; Diphtheria | interventions — adacel; Diphtheria-Tetanus Vaccine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Adacel Vaccine Group (Experimental)
  Interventions: Biological: ADACEL®: Tetanus, Reduced Diphtheria and Acellular Pertussis Adsorbed
- DECAVAC Vaccine Group (Active Comparator)
  Interventions: Biological: DECAVAC®: Tetanus and Diphtheria Toxoids Adsorbed

INTERVENTIONS:
Biological: ADACEL®: Tetanus, Reduced Diphtheria and Acellular Pertussis Adsorbed — 0.5 mL, IM
  Other Names: ADACEL®
  Arms: Adacel Vaccine Group
Biological: DECAVAC®: Tetanus and Diphtheria Toxoids Adsorbed — 0.5 mL, IM
  Other Names: DECAVAC®
  Arms: DECAVAC Vaccine Group

SUMMARY:
It is well recognized that older adults can contract pertussis, suffer its complications, and unwittingly transmit it to close contacts, which may well include infants too young to have received their primary series of DTaP vaccinations. ADACEL® vaccine is currently licensed in the US for persons 11 - 64 years of age, but no pertussis vaccine is yet approved for administration to older adults. The most widely used Td vaccine in the US, DECAVAC®, has no upper limit on its age indication.

The purpose of this trial is to describe the safety and immunogenicity of ADACEL® vaccine among individuals ≥ 65 years of age.

ELIGIBILITY:
Inclusion Criteria :

* Ambulatory and not institutionalized.
* At least 65 years of age at the time of vaccination.
* Signed Institutional Review Board (IRB)-approved informed consent form.
* Able to attend all scheduled visits and to comply with all trial procedures.

Exclusion Criteria :

* Any condition which, in the opinion of the investigator, would pose a health risk to the participant or interfere with the evaluation of the vaccine.
* Serious chronic disease (eg, cardiac, renal, neurologic, metabolic, rheumatologic, psychiatric) that is unstable or that, in the opinion of the investigator, might:

  * interfere with the ability to participate fully in the study; or
  * interfere with evaluation of the vaccine.
* Known or suspected impairment of immunologic function, including use of immune suppressive medications (eg, rheumatoid arthritis drugs such as methotrexate; cancer chemotherapy agents such as vincristine).
* Febrile illness within the last 72 hours or an oral temperature ≥ 100.4°F (≥ 38°C) at the time of inclusion.
* Any history of documented tetanus, diphtheria or pertussis disease.
* Known or suspected receipt of a tetanus, diphtheria or acellular pertussis containing vaccine within the preceding 5 years.
* Administration of immune globulin or other blood products within the last three months, or systemic corticosteroid therapy (prednisone or equivalent) for more than 2 consecutive weeks within the past 6 months.
* Systemic antibiotic therapy within the 72 hours prior to enrollment.
* Received any vaccine, other than influenza vaccine, in the 30-day period prior to enrollment or scheduled to receive any vaccine, other than influenza vaccine, in the 35-day period after enrollment. For influenza vaccine only, defer if received in the 14-day period prior to enrollment or scheduled to receive in the 14-day period after enrollment.
* Suspected or known hypersensitivity to any of the vaccine components.
* Participation in another interventional clinical trial in the 4 weeks preceding enrollment or planning to participate in another interventional clinical trial during the planned period of this study.
* Use of alcohol or drugs in a manner that may, in the opinion of the investigator, interfere with the subject's ability to comply with trial visits or procedures.
* Thrombocytopenia or bleeding disorder contraindicating intramuscular vaccination.
* Subject deprived of freedom by an administrative or court order, or in an emergency setting, or hospitalized without his/her consent, or requires a legally authorized representative.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 1564 (Actual)
Dates: Start 2007-03; Primary Completion 2008-09 (Actual); Study Completion 2008-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Sanofi Pasteur Inc.
Locations (18):
- United States (18):
  - Chandler, Arizona
  - Phoenix, Arizona
  - Cypress, California
  - San Luis Obispo, California
  - Atlanta, Georgia
  - Chicago, Illinois
  - New Orleans, Louisiana
  - Rockville, Maryland
  - Minneapolis, Minnesota
  - St Louis, Missouri
  - Akron, Ohio
  - Cincinnati, Ohio
  - Mogadore, Ohio
  - Knoxville, Tennessee
  - Salt Lake City, Utah
  - West Jordan, Utah
  - Annandale, Virginia
  - Williamsburg, Virginia

REFERENCES:
- See also: Related Info — http://www.sanofipasteur.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled from 28 March to 30 October 2007, at 19 clinic centers in United States.
Pre-assignment Details: A total of 1563 participants were enrolled; 1561 were vaccinated with data analyzed and presented in this report.
Groups:
- ADACEL® Vaccine Group: Participants received a single dose of ADACEL® vaccine.
- DECAVAC® Vaccine Group: Participants received a single dose of DECAVAC® vaccine.
Period: Overall Study
Arm/Group | ADACEL® Vaccine Group | DECAVAC® Vaccine Group
Started | 1170 | 391
Completed | 1158 | 389
Not Completed | 12 | 2
Not completed — Lost to Follow-up | 3 | 0
Not completed — Protocol Violation | 4 | 1
Not completed — Withdrawal by Subject | 3 | 1
Not completed — Serious Adverse Events | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- DECAVAC® Vaccine Group: Participants received a single dose of ADACEL® vaccine.
- Total: Total of all reporting groups
Arm/Group | ADACEL® Vaccine Group | DECAVAC® Vaccine Group | Total
Number analyzed (Participants) | 1170 | 391 | 1561
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 1170 | 391 | 1561
Age Continuous [Mean (Standard Deviation); unit: Years] | 72.2 (5.74) | 72.3 (5.63) | 72.2 (5.71)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 579 | 198 | 777
  Male | 591 | 193 | 784
Region of Enrollment [Number; unit: participants]
  United States | 1170 | 391 | 1561

OUTCOME MEASURES:

1. Primary Outcome: Geometric Mean Titers (GMTs) of Tetanus, Diphtheria, and Pertussis Antibodies Pre- and Post-Vaccination With ADACEL® or DECAVAC® Vaccine
Time Frame: Day 35 post-vaccination
Population: GMTs and their 95% Confidence Intervals were assessed in the per-protocol population.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | ADACEL® Vaccine Group | DECAVAC® Vaccine Group
Number analyzed (Participants) | 1094 | 371
Titers
  Tetanus (Pre-vaccination: N = 1089; 368) | 0.501 [0.445 to 0.564] | 0.451 [0.365 to 0.558]
  Tetanus (Post-vaccination: N = 1075; 368) | 8.43 [7.78 to 9.14] | 7.23 [6.23 to 8.38]
  Diphtheria (Pre-vaccination: N = 1092; 370) | 0.049 [0.043 to 0.056] | 0.056 [0.045 to 0.071]
  Diphtheria (Post-vaccination: N = 1093; 371) | 0.570 [0.489 to 0.665] | 0.505 [0.401 to 0.636]
  Pertussis Toxoid (Pre-vaccination: N = 1013; 345) | 10.6 [9.81 to 11.5] | 12.7 [11.1 to 14.5]
  Pertussis Toxoid (Post-vaccination: N = 1022; 341) | 59.4 [55.2 to 63.8] | 15 [13.1 to 17.2]
  Filamentous Hemagglutinin (Pre-vacc: N=1091; 370) | 25.5 [23.9 to 27.1] | 25.6 [22.8 to 28.8]
  Filamentous Hemagglutinin (Post-Vacc: N=1094; 371) | 197 [186 to 209] | 26.6 [23.7 to 30]
  Pertactin (Pre-Vaccination: N = 1090; 370) | 4.56 [4.26 to 4.88] | 4.71 [4.18 to 5.31]
  Pertactin (Post-Vaccination: N = 1094; 370) | 69.2 [61.6 to 77.9] | 5.34 [4.72 to 6.04]
  Fimbriae Type 2 & 3 (Pre-Vaccination: N=1053; 370) | 8.28 [7.46 to 9.19] | 9.59 [7.94 to 11.6]
  Fimbriae Type 2 & 3 (Post-Vaccination: N=1060; 352 | 183 [164 to 205] | 10.6 [8.79 to 12.9]

2. Primary Outcome: Percentage of Participants With Post-vaccination Tetanus and Diphtheria Concentrations ≥0.10 IU/mL (Seroprotection) ADACEL® or DECAVAC®.
Description: Seroprotection was defined as a post-vaccination Concentrations of ≥0.10 IU/mL.
Time Frame: Day 35 post-vaccination
Population: Seroprotection was assessed in the per-protocol population
Measure: Number; unit: Percentage of Participants
Arm/Group | Adacel® Vaccine Group | DECAVAC® Vaccine Group
Number analyzed (Participants) | 1093 | 371
Percentage of Participants
  Tetanus (N = 1075; 368) | 98 | 98
  Diphtheria (N = 1093; 371) | 77 | 79

3. Primary Outcome: Percentage of Participants With Booster Response to Tetanus and Diphtheria Post-vaccination With ADACEL® or DECAVAC® Vaccine.
Description: Booster response was defined as a minimum rise in antibody concentration from pre- to post-vaccination. The minimum rise is at least 2 times, if pre-vaccination concentration is above the the cutoff value (Tetanus 5.47 IU/mL; Diphtheria 1.28 IU/mL) or at least 4 times it it is at or below the cutoff value.
Time Frame: Day 35 post-vaccination
Population: Booster response was assessed in the per-protocol population.
Measure: Number; unit: Percentage of Participants
Arm/Group | ADACEL® Vaccine Group | DECAVAC® Vaccine Group
Number analyzed (Participants) | 1091 | 370
Percentage of Participants
  Tetanus (N = 1071; 365) | 77 | 77
  Diphtheria (N = 1091; 370) | 71 | 66

4. Other Pre Specified Outcome: Number of Participants With At Least One Solicited Injection Site or Systemic Reaction Post-vaccination With Either ADACEL® or DECAVAC® Vaccine.
Description: Solicited injection site reactions: Pain, Erythema, and Swelling; Solicited systemic reactions; Fever (Temperature), Headache, Myalgia, and Malaise.
Time Frame: Day 0 up to 14 days post-vaccination
Population: Safety analysis was on all enrolled and vaccinated participants, intend-to-treat population.
Measure: Number; unit: Participants
Arm/Group | ADACEL® Vaccine Group | DECAVAC® Vaccine Group
Number analyzed (Participants) | 1170 | 391
Participants
  Any Solicited Injection Site Reaction | 615 | 200
  Any injection site Pain | 496 | 163
  Grade 3 injection site Pain (Incapacitating) | 6 | 1
  Any injection site Erythema | 280 | 86
  Grade 3 injection site Erythema (≥ 3.5 cm) | 52 | 19
  Any injection site Swelling | 209 | 59
  Grade 3 injection site Swelling (≥ 3.5 cm) | 40 | 17
  Any Solicited Systemic Reaction | 420 | 155
  Any Fever | 6 | 2
  Grade 3 Fever (≥ 39.5ºC or ≥ 103.1ºF) | 1 | 0
  Any Headache | 209 | 76
  Grade 3 Headache (Incapacitating) | 7 | 4
  Any Myalgia | 327 | 108
  Grade 3 Myalgia (Incapacitating) | 17 | 6
  Any Malaise | 198 | 63
  Grade 3 Malaise (Incapacitating) | 13 | 6

ADVERSE EVENTS:
Time Frame: Adverse events data were collected from the day of vaccination (Day 0) for up to 6 months post-vaccination.
Arm/Group | ADACEL® Vaccine Group | DECAVAC® Vaccine Group
Serious Adverse Events (participants affected / at risk) | 49/1170 | 20/391
Other Adverse Events (participants affected / at risk) | 615/1170 | 200/391
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ADACEL® Vaccine Group (N=1170) | DECAVAC® Vaccine Group (N=391)
Acute coronary syndrome (Cardiac disorders) | 0 (0) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Arrhythmia (Cardiac disorders) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 4 (4) | 0 (0)
Cardiac arrest (Cardiac disorders) | 1 (1) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 4 (4) | 1 (1)
Coronary artery disease (Cardiac disorders) | 3 (3) | 1 (1)
Intracardiac thrombus (Cardiac disorders) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 2 (2) | 0 (0)
Adrenocortical insufficiency chronic (Endocrine disorders) | 1 (1) | 0 (0)
Barrett's oesophagus (Gastrointestinal disorders) | 1 (1) | 0 (0)
Duodenal ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Melaena (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Volvulus (Gastrointestinal disorders) | 1 (1) | 0 (0)
Adverse drug reaction (General disorders) | 0 (0) | 1 (1)
Hernia obstructive (General disorders) | 1 (1) | 0 (0)
Multi-organ failure (General disorders) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 1 (1) | 0 (0)
Bile duct stone (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 2 (2) | 2 (2)
Appendicitis (Infections and infestations) | 1 (1) | 2 (2)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0)
Bursitis infective (Infections and infestations) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1)
Diverticulitis (Infections and infestations) | 0 (0) | 1 (1)
Escherichia infection (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 3 (3) | 1 (1)
Sepsis (Infections and infestations) | 2 (2) | 0 (0)
Staphylococcal bacteraemia (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1)
Viral infection (Infections and infestations) | 1 (1) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Joint injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Meniscus lesion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Spinal fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Stent occlusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Diabetes mellitus non-insulin-dependent (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Muscle haemorrhage (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Myositis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Hepatic neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Renal cell carcinoma stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Small cell lung cancer stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Uterine cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 4 (4) | 1 (1)
Intracranial venous sinus thrombosis (Nervous system disorders) | 1 (1) | 0 (0)
Subarachnoid haemorrhage (Nervous system disorders) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 1 (1) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 1 (1) | 1 (1)
Hydronephrosis (Renal and urinary disorders) | 2 (2) | 0 (0)
Renal artery stenosis (Renal and urinary disorders) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 1 (2)
Hypertensive crisis (Vascular disorders) | 1 (1) | 0 (0)
Peripheral embolism (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | ADACEL® Vaccine Group (N=1170) | DECAVAC® Vaccine Group (N=391)
Injection site pain (General disorders) | 496 | 163
Injection site erythema (General disorders) | 280 | 86
Injection site swelling (General disorders) | 209 | 59
Headache (Nervous system disorders) | 209 | 76
Myalgia (Musculoskeletal and connective tissue disorders) | 327 | 108
Malaise (General disorders) | 198 | 63

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor must have the opportunity to review at least 60 days prior to submission for publication or presentation. If review indicates that potentially patentable subject matter would be disclosed, publication or public disclosure may be delayed for a maximum of an additional 60 days to allow for filing the necessary patent applications.